CLINICAL TRIAL: NCT05404841
Title: Investigating the Effect of Whole-fruit Coffee Extract on Exercise Performance
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: VDF FutureCeuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-10-20-B-05
Record Dates: First submitted 2022-01-10; First posted 2022-06-03 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Caffine and Endurance Performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CoffeeBerry Supplement (Experimental): Caffeine and polyphenol supplement
  Interventions: Dietary Supplement: CoffeeBerry Supplement
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CoffeeBerry Supplement — A Coffeeberry supplement containing 200mg Caffeine and 14mg polyphenols, manufactured by FutureCeuticals Inc.,
  Arms: CoffeeBerry Supplement
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Caffeine is a widely used efficacious supplement by both the general public, and athletes, with the goal of improving performance. The effects of caffeine alone are well known, but it is not clear whether a multi-ingredient supplement (containing both caffeine and polyphenols) can affect exercise performance.

This study aims to determine if a low dose of caffeine, in the form of a whole-fruit coffee extract also containing polyphenols, can improve exercise performance compared to a placebo condition, with a secondary objective of identifying if this supplement can improve post exercise refuelling (glycogen resynthesis).

Participants will consume either the supplement or a placebo before engaging in an exercise protocol. Muscle biopsies will then be obtained so as to measure subsequent glycogen resynthesis, with multiple blood samples being taken through the day. The following morning another biopsy will be taken before the exercise protocol will be repeated.

This research will inform us of the efficacy of caffeine and polyphenols on improving exercise performance.

ELIGIBILITY:
Exclusion criteria:

* Allergy to Lidocaine
* Exclusion critera
* Any diagnosed metabolic health condition
* Pregnant
* Non-habitual caffeine intake
* Smoker
* No endurance training
* Diagnosed Cardiovascular disease
* Beta-Blockers
* Recent history of musculoskeletal injury

Inclusion criteria:

* Age 18-40
* Heathy
* Highly trained endurance athletes (V̇O2max: males >55 and females >50 mL⋅kg bm-1⋅min-1)
* Both males and females are allowed to participate. If females are on the oral contraceptive pill they are to be tested on consecutive weeks. If they are not on the oral contraceptive pill, then female subjects are to be tested every 4 weeks, at the same point of their menstrual cycle.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Exercise performance | 15 Minitues
  Amount of work completed in 15 minutes

SECONDARY OUTCOMES:
Glycogen Resynthesis | 24 Hours
  The diffrence in glycogen within the muscle between two time points
Alertness | 1 Minitue
  10 cm visual analog scale (Ranging from Not Alert to Extremly Alert)
Motivation | 1 Minitue
  10 cm visual analog scale (Ranging from Not motivated to Extremly motivated)
Rate of perceived exertion | 1 Minitue
  Validated Borg scale (6-20 Arbitrary units)
Urine osmolarity | 24 Hours
  The hydration status of the individual measured in mOsmo|/kg
GI comfort | 1 Minitue
  10 cm visual analog scale (Ranging from No discomfort to Extreme discomfort)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Sport & Health Sciences University of Exeter, Exeter, Devon
  - University of Exeter, Exeter

IPD SHARING:
Plan to Share IPD: No